CLINICAL TRIAL: NCT02351674
Title: A Single Centre, Retrospective Cohort Study on Post Analysis on the Link Between the Clinical Heart Rate and Outcomes During PCI
Brief Title: Retrospective Cohort Study on Post Analysis on the Link Between the Clinical Heart Rate and Outcomes During PCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dandan Li (Other)
Responsible Party: Sponsor-Investigator, Dandan Li, M.D., Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: ESR-14-10413
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Coronary Heart Disease
Keywords: Heart Rate; Percutaneous coronary intervention; outcome
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Heart rate ≤70bpm: 15,000 patients in the retrospective cohort will be divided into 4 groups according to their mean heart rate during PCI. Group 1 will be defined as subjects' mean heart rate ≤70 BPM.
- Heart rate between 71 to 80bpm: 15,000 patients in the retrospective cohort will be divided into 4 groups according to their mean heart rate during PCI. Group 2 will be defined as subjects' mean heart rate between 71 to 80bpm.
- Heart rate between 81 to 90bpm: 15,000 patients in the retrospective cohort will be divided into 4 groups according to their mean heart rate during PCI. Group 1 will be defined as subjects' mean heart rate between 81 to 90bpm.
- Heart rate>90bpm: 15,000 patients in the retrospective cohort will be divided into 4 groups according to their mean heart rate during PCI. Group 4 will be defined as subjects' mean heart rate>90bpm

SUMMARY:
The trial is a single centre, retrospective cohort, non-interventional study to be conducted in the department of cardiology, Chinese PLA General Hospital, Beijing, China. To evaluate the link between mean perioperative clinical heart rate and short-term composite outcomes during PCI among local CHD patients.

DETAILED DESCRIPTION:
The study requires those data including subjects aged from 20 to 80 year-old, diagnosed as coronary heart disease with records on mean clinical heart rate during PCI from 2009.1 to 2014.5 in the database from the department of cardiology, Chinese PLA General Hospital, Beijing. All 15,000 subjects' related data from the database will be collected.Once selected, 15,000 patients in the retrospective cohort will be divided into 4 groups according to their mean clinical resting heart rate during PCI. Group 1 will be defined as subjects' mean clinical resting heart rate ≤70 BPM, which will be set as baseline. Group 2 will be defined as subjects' mean clinical resting heart rate between 71 to 80 BPM. Group 3 will be defined as subjects' mean clinical resting heart rate between 81 to 90 BPM. Group 4 will be defined as subjects' mean clinical resting heart rate >90 BPM. The primary endpoint is to determine the link between the mean perioperative heart rate and short-term outcomes during PCI among local CHD patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients consecutive enrolled in Chinese PLA General Hospital from January 2009 to May 2014
* Diagnosed as coronary heart disease with records on mean clinical heart rate during PCI .

Exclusion Criteria:

* Inferior wall myocardial infarction (MI) history or/and acute inferior wall MI patients;
* Dead within 3 days after admit into wards;
* LVEF<30%;
* Install a permanent pacemaker patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study requires those data including subjects aged from 20 to 80 year-old, diagnosed as coronary heart disease with records on mean clinical heart rate during PCI from 2009.1 to 2014.5 in the database from the department of cardiology, Chinese PLA General Hospital, Beijing.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with composite events including CVD mortality, fatal/non-fatal MI, non-fatal sudden cardiac arrest, fatal/non-fatal stroke and malignant arrhythmia | During PCI

SECONDARY OUTCOMES:
Mean perioperative clinical heart rate | During PCI
  The primary efficacy endpoint is proportion of patients with composite events including CVD mortality, fatal/non-fatal MI, non-fatal sudden cardiac arrest, fatal/non-fatal stroke and malignant arrhythmia.
Clinical resting heart rate and heart rate variability | During PCI

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Ph.D., Principal Investigator — Ph.D. advisor

REFERENCES:
- [Background] Fox K, Borer JS, Camm AJ, Danchin N, Ferrari R, Lopez Sendon JL, Steg PG, Tardif JC, Tavazzi L, Tendera M; Heart Rate Working Group. Resting heart rate in cardiovascular disease. J Am Coll Cardiol. 2007 Aug 28;50(9):823-30. doi: 10.1016/j.jacc.2007.04.079. Epub 2007 Aug 13. PMID 17719466
- [Background] Ho JE, Bittner V, Demicco DA, Breazna A, Deedwania PC, Waters DD. Usefulness of heart rate at rest as a predictor of mortality, hospitalization for heart failure, myocardial infarction, and stroke in patients with stable coronary heart disease (Data from the Treating to New Targets [TNT] trial). Am J Cardiol. 2010 Apr 1;105(7):905-11. doi: 10.1016/j.amjcard.2009.11.035. PMID 20346304
- [Background] Kolloch R, Legler UF, Champion A, Cooper-Dehoff RM, Handberg E, Zhou Q, Pepine CJ. Impact of resting heart rate on outcomes in hypertensive patients with coronary artery disease: findings from the INternational VErapamil-SR/trandolapril STudy (INVEST). Eur Heart J. 2008 May;29(10):1327-34. doi: 10.1093/eurheartj/ehn123. Epub 2008 Mar 29. PMID 18375982
- [Background] Anselmino M, Ohrvik J, Ryden L; Euro Heart Survey Investigators. Resting heart rate in patients with stable coronary artery disease and diabetes: a report from the euro heart survey on diabetes and the heart. Eur Heart J. 2010 Dec;31(24):3040-5. doi: 10.1093/eurheartj/ehq368. Epub 2010 Oct 8. PMID 20935002